CLINICAL TRIAL: NCT02442609
Title: Does Patient Look to Internet for Anesthesia Information Before Surgery : a Prospective International Questionaire Study
Brief Title: Internet for Anesthesia Information : a Patient Questionaire
Acronym: e-anesth
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Philippe Cuvillon, MD, PhD, Pierre and Marie Curie University
Other Study IDs: PMCurrieU
Record Dates: First submitted 2015-05-09; First posted 2015-05-13 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Anaesthesia
Keywords: internet; anesthesia; information; surgery; question

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patient: patient schedulled for elective surgery, adult (> 18yrs), non emergency procedure, able to read questionaire
  Interventions: Other: questionaire

INTERVENTIONS:
Other: questionaire — questionaire before surgery

SUMMARY:
Patients need information for perioperative period and internet may be an interesting alternative.This study analysed by questionaire what does patient look on internet: information of perioperative period and specifically for anesthesia. Questionaire (8 questions) are distributed to the patient before surgery and after they were prepared by surgeon. Population : adult (> 18 y), no emergency procedure.The mean question is the use of internet for anesthesia information.

DETAILED DESCRIPTION:
This is a prospective study with 23 centers ( France, Suisse, Belgium, Canada) including before surgery: adult (> 18y), no emergency procedure. Questionaires (8 questions) are distributed to the patient before surgery and after they were prepared by surgeon. After collecting all questionaires, questionaires are analysed by an independant center. The mean question is the use of internet for anesthesia information. More than 8000 patients have to be enrolled during the study period over 23 centers.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 yr)
* surgery
* private or public hospital

Exclusion Criteria:

* refusal,
* emergency surgery
* epidural analgesia for pregnant patient

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (> 18 yrs), schedulled for surgery under local, regional or general surgery
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
use of internet | 1 day
  response to the question: yes or not

SECONDARY OUTCOMES:
Age | 1 day
  age, type of surgery
search of anesthesia informations | 1 day
  questions to know what patient are loocking for
social activity | 1 day
  active or not
surgery | 1 day
  type of surgery for patient
interest for pre operative questionaire for anesthesia | 1 day
  yes vs no

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Leclerc, MD, Principal Investigator — ICM, CRLC, Montpellier, France; Philippe Cuvillon, MD, PhD, Study Director — ICM, CRLC, Montpellier, France
Locations (2):
- France (2):
  - CHU Caremeau, Nîmes, GArd
  - CHU Toulouse, Toulouse

REFERENCES:
- [Derived] Nucci B, Claret PG, Leclerc G, Chaumeron A, Grillo P, Buleon C, Leprince V, Raux M, Minville V, Futier E, Lefrant JY, Cuvillon P; Anaesthesia Internet Study Group. Role of the internet as an information resource before anaesthesia consultation: A French prospective multicentre survey. Eur J Anaesthesiol. 2017 Dec;34(12):831-835. doi: 10.1097/EJA.0000000000000686. PMID 28922337